CLINICAL TRIAL: NCT05566834
Title: A Phase 1 Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Minnelide™ Capsules Given Alone or in Combination With Paclitaxel in Patients With Advanced Gastric Cancer
Brief Title: Minnelide™ Capsules Alone and in Combination With Paclitaxel in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneamrita Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minnelide GC 101
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — 14-O-phosphonooxymethyltriptolide disodium salt

STUDY DESIGN:
Intervention Model Description: Minnelide™ is a water soluble disodium salt variant of triptolide, a diterpenoid, an HSP70 inhibitor. Studies using orthotopic pancreatic cancer cell lines and human xenograft transplants demonstrate that Minnelide™ prevents tumor progression, increases survival, and causes tumor regression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label, dose-escalation, safety, Pharmacodynamic, pharmacokinetic study. (Experimental): One
  Interventions: Drug: Minnelide

INTERVENTIONS:
Drug: Minnelide — at the MTD dose level established for monotherapy or combination to confirm safety. With a sample of 12 patients, the probability is > 80% that a serious adverse event with at least a 16% incidence will be detected.

SUMMARY:
A Phase 1, Open-label, Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of Minnelide™ Capsules given alone or in combination with paclitaxel in patients with Advanced Gastric Cancer.

DETAILED DESCRIPTION:
Minnelide™ is a water soluble disodium salt variant of triptolide, a diterpenoid, an HSP70 inhibitor. Studies using orthotopic pancreatic cancer cell lines and human xenograft transplants demonstrate that Minnelide™ prevents tumor progression, increases survival, and causes tumor regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced gastric cancer

  * Tumor progression after receiving standard/approved chemotherapy or where there is no approved therapy
  * One or more metastatic tumors measurable per RECIST v1.1 Criteria
  * Karnofsky performance ≥ 70%
  * Life expectancy of at least 3 months
  * Age ³ 19 years
  * Signed, written IRB-approved informed consent
  * A negative pregnancy test (if female)
  * Acceptable liver function:

    * Bilirubin 1.5 times upper limit of normal
    * AST (SGOT), ALT (SGPT) and Alkaline phosphatase 2.5 times upper limit of normal (if liver metastases are present, then 5 x ULN is allowed)
    * Albumin ≥ 3.0 g/dL
  * Acceptable renal function:

    o Serum creatinine within normal limits, OR calculated creatinine clearance ³ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * Acceptable hematologic status:

    * Granulocyte

      * Monotherapy: ³ 1,500 cells/mm3
      * Combination therapy with paclitaxel: ³ 2,000cells/mm3 Platelet count ³ 100,000 (plt/mm3)
    * Hemoglobin ³ 9 g/dL
  * Urinalysis:

    o No clinically significant abnormalities
  * Acceptable coagulation status:

    * PT ≤ 1.5 times institutional ULN
    * PTT ≤ 1.5 times institutional ULN
  * Women of child- bearing potential and men must agree to use adequate contraception For men and women of child-producing potential, the use of effective contraceptive methods during the study and until 90 days after the last dose of IP for men or until 6 months after the last dose of IP for women or 6 months after the last dose of IP with paclitaxel for both men and women.

Exclusion Criteria:

New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG

* Baseline QTc exceeding 470 msec (using the Bazett's formula) and/or patients receiving class 1A or class III antiarrhythmic agents.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Pregnant or nursing women. NOTE: For men and women of child-producing potential, the use of effective contraceptive methods during the study and until 90 days after the last dose of IP for men or until 6 months after the last dose of IP for women or 6 months after the last dose of IP with paclitaxel for both men and women. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Treatment with radiation therapy (local therapy, non-target lesion, 2 weeks), major surgery, chemotherapy, biological agents or investigational therapy within 3 weeks prior to study treatment.
* Unwillingness or inability to comply with procedures required in this protocol
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent
* Patients who are on a prohibited medication (section 4.3.2).
* Patients with biliary obstruction and/or biliary stent (Regimen B only)
* Patients with a history of severe hypersensitivity reactions to products containing Cremophor® EL (eg, cyclosporin for injection concentrate and teniposide for injection concentrate). • Patient with baseline ANC<1500/mm3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To determine any increase of treatment emergent adverse events when Minnelide capsules are given in combination with paclitaxel. | 24 months
  To observe any increase in the number of patients that experience Grade 4 neutropenia lasting ≥ 5 days or Grade 3 or 4 neutropenia with fever and/or infection; Grade 4 thrombocytopenia (or Grade 3 with bleeding); Grade 3 or 4 treatment-related non-hematological toxicity (Grade 3 nausea, vomiting or diarrhea that last > 72 hours despite maximal treatment when Minnelide is given alone and in combination with paclitaxel compared to the incidence with gemcitabine and nab-paclitaxel.

SECONDARY OUTCOMES:
Pharmacokinetics of Minnelide when given with paclitaxel | 24 months
  Area under the concentration curve (AUC) will be determine the exposure of Minnelide
Plasma levels of Minnelide when given with paclitaxel | 24 months
  Maximum plasma concentration (Cmax) will be measured to determine the effect of Minnelide when given with paclitaxel

CONTACTS AND LOCATIONS:
Overall Officials: Mohana Velagapudi, Study Director — Minneamrita Therapeutics LLC
Locations (1):
- Samsung Medical Center, Soeul, South Korea

IPD SHARING:
Plan to Share IPD: No